CLINICAL TRIAL: NCT00859976
Title: Prospective Randomised Control Trial to Compare the Effect Upon Bone Density and Clinical Outcomes When Using BoneMaster HA Coated Acetabular Cups Compared With Plasma Sprayed HA Coated Cups in Patients With Total Hip Replacements
Brief Title: Study Comparing BoneMaster Hydroxyapatite Coating With Plasma-sprayed Hydroxyapatite Coating on Acetabular Cups
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMETEU.CR.EU27; UK REC Ref: 08/H0724/24
Record Dates: First submitted 2009-03-06; First posted 2009-03-11 (Estimated); Results first posted 2019-02-08 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Arthropathy of Hip
Keywords: BoneMaster; Total Hip Replacement; Bone Density; Patients suitable for Total Hip Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Plasma-sprayed shell (Active Comparator): Exceed ABT plasma-sprayed hydroxyapatite coated acetabular cup.
  Interventions: Device: Plasma Coated Acetabular Shell
- BoneMaster coated shell (Experimental): Exceed ABT BoneMaster hydroxyapatite coated acetabular cup.
  Interventions: Device: BoneMaster coated acetabular shell.

INTERVENTIONS:
Device: BoneMaster coated acetabular shell. — Bonemaster coated Exceed Acetabular Shell
  Other Names: Bonemaster coated Exceed Acetabular Shell
  Arms: BoneMaster coated shell
Device: Plasma Coated Acetabular Shell — Plasma HA coated Exceed Acetabular Shell
  Other Names: Plasma Hydroxyapatite coated Exceed Acetabular Shell
  Arms: Plasma-sprayed shell

SUMMARY:
The randomised controlled trial will be carried out on patients that require a total hip replacement (THR) to reduce pain and restore their function. One way of fixing the hip joint to the bone is by coating the implant to encourage the body to grow bone onto the replacement hip. This study is aiming to find out whether the new (Bonemaster) coating allows increased bony growth onto the cup when compared to the usual (plasma-sprayed) coating. This may reduce the incidence of early failures due to poor bony attachment, which is a well known complication for early failure of total hip replacements.

The study will compare two different types of coating (BoneMaster and Plasma-sprayed) on the cup of the replacement hip. Density of the bone immediately surrounding the cup will be observed to see if there are differences between the two groups. The density of bone will be measured using standard x-ray assessment and in a smaller sample of 14 patients, using a special scan called Dual Energy X-ray Absorptiometry (DEXA Scan). Functional comparisons will be assessed through clinical scores.

DETAILED DESCRIPTION:
The patients will be identified by the orthopaedic surgeon in the orthopaedic clinic and deemed suitable for the study if all inclusion and exclusion criteria are met. 210 patients will be recruited to the study and each patient will be randomised into either of the groups allowing 105 patients into each group. Patients will be followed up at 6 months, 1 year and 2 years after the surgery. All patients will have radiographic assessments at these follow-up intervals, as well as Harris Hip, Oxford Hip and Womac scores. This will allow comparison of the two groups.

The BoneMaster coating has been extensively tested in cell and animal studies and has been evaluated in one previous clinical study and showed favorable results. Further investigation is required to ensure the new coating may enhance bony growth allowing better fixation of the hips in the early period after the operation and also over a longer period of time. The growth needs to be measured using a more sensitive scan than radiographic assessment alone, called DEXA which was also used in the previous study.

ELIGIBILITY:
Inclusion Criteria

* Patients suitable for THR surgery with a diagnosis of Osteoarthritis
* Patients aged 40 -85 years old.
* Patients with limited co-morbidity - ASA I - III (low risk for surgery)
* Patients must be able to understand instructions and be willing to return for follow up

Exclusion Criteria

* Rheumatoid arthritis
* Patients requiring supplemental screw fixation
* Previous hip surgery to the affected hip
* Patients with significant co-morbidity - ASA IV - V (high risk for surgery)
* Dementia
* Neurological conditions affecting everyday functional ability and hip movement
* The patient is unable to give informed consent
* Patients who have suffered from cancer
* The patient is currently part of another research study
* Patients who need to take Non Steroidal Anti-inflammatory Drugs (NSAIDs) in the first 6 weeks after surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2009-03; Primary Completion 2012-06 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helmut ZAHN, Principal Investigator — William Harvey Hospital
Locations (1):
- William Harvey Hospital, Ashford, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Plasma-sprayed Shell | BoneMaster Coated Shell
Started | 82 | 85
Completed | 66 | 67
Not Completed | 16 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Plasma-sprayed Shell | BoneMaster Coated Shell | Total
Number analyzed (Participants) | 82 | 85 | 167
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (7) | 70 (9) | 68.55 (8.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 51 | 94
  Male | 39 | 34 | 73

OUTCOME MEASURES:

1. Primary Outcome: Record and Measure Bone Density Using DEXA Scans at 24 Months.
Description: DEXA scan cohort - DEXA scan was used to measure bone density. Below is the calculated net average bone mineral density (BMD) percentage change from baseline at 2 years.
Time Frame: 2 years.
Population: DEXA scan cohort: Bonemaster group, n = 7; Plasma-Sprayed group, n = 7
Measure: Mean (Standard Deviation); unit: Net average BMD %change from baseline
Arm/Group | Plasma-sprayed Shell | BoneMaster Coated Shell
Number analyzed (Participants) | 7 | 7
Net average BMD %change from baseline | -11.0 (4.0) | 5.7 (57.3)
Statistical Analysis 1: Comparison: Plasma-sprayed Shell vs BoneMaster Coated Shell; Test type: Superiority — A superiority test was used to calculate the number of patients that are needed in order to show a difference between the bone mineral density surrounding BoneMaster coated cups compared to plasma HA sprayed cups; p = 0.4570, Wilcoxon (Mann-Whitney); Change in bone mineral density, normalised to baseline levels

2. Secondary Outcome: Secondary Outcomes Are Functional Assessment Using Harris Hip Score
Description: Modified Harris Hip Score, total score 0-100. A score of <70 is poor, 70-79 is fair, 80-89 is good, 90-100 is excellent.
Time Frame: 2 years
Population: 2 years post-op
Measure: Least Squares Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Plasma-sprayed Shell | BoneMaster Coated Shell
Number analyzed (Participants) | 59 | 60
Units on a scale | 83.92 (15.82) | 81.83 (20.79)

3. Secondary Outcome: Secondary Outcomes Are Clinical Assessment Using Oxford Hip Score
Description: Oxford Hip Score, scored 12-60. The Oxford hip score - this score was based on the original publication where each answer gives a score of 1-5. A score of 1 for each question, represented best outcome/least symptoms. Therefore a total score of 12 was the best overall outcome.
Time Frame: 2 years.
Population: 2 years post-op
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Plasma-sprayed Shell | BoneMaster Coated Shell
Number analyzed (Participants) | 59 | 61
Units on a scale | 19.2 (8) | 19.8 (9.2)

4. Secondary Outcome: Secondary Outcomes Are Clinical Assessment Using WOMAC Hip Score
Description: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Hip Score, Each question is scored on a scale of 0 (best health state) to 4 (worst health state); total WOMAC hip score, 0 being the best and 96 being the worst.
Time Frame: 2 years
Population: 2 years post-op
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Plasma-sprayed Shell | BoneMaster Coated Shell
Number analyzed (Participants) | 41 | 47
Units on a Scale | 14.2 (16.5) | 12.1 (17.4)

5. Primary Outcome: Radiography to Determine Radiolucency in All Three DeLee & Charnley Zones of the Acetabulum.
Description: 34 patient cases without duplicated data were the basis for the radiographic analysis that was conducted: Bonemaster group, n = 12; Plasma-Sprayed group, n = 22. The degree of osseous-fixation was determined by grading: 1-2 mm radiolucencies, classed as not fixated; >2mm radiolucencies, classed as unstable.
Time Frame: 2 years.
Measure: Count of Participants; unit: Participants
Arm/Group | Plasma-sprayed Shell | BoneMaster Coated Shell
Number analyzed (Participants) | 22 | 12
Participants
  1-2 mm radiolucency in Zone B1 | 3 | 0
  >2 mm radiolucency in zone B2 | 1 | 0

ADVERSE EVENTS:
Arm/Group | Plasma-sprayed Shell | BoneMaster Coated Shell
Serious Adverse Events (participants affected / at risk) | 1/82 | 2/85
Other Adverse Events (participants affected / at risk) | 5/82 | 10/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Plasma-sprayed Shell (N=82) | BoneMaster Coated Shell (N=85)
Death (General disorders) | 0 | 2 — Patient Deaths that were reported over the course of the study; considered SAE
Dislocation (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Plasma-sprayed Shell (N=82) | BoneMaster Coated Shell (N=85)
Cardiovascular - stroke (Cardiac disorders) | 0 | 1
Fractured pelvis (Musculoskeletal and connective tissue disorders) | 0 | 1
Fall - patient confused (General disorders) | 0 | 2
Urogenital adverse event with diarrhoea (Renal and urinary disorders) | 0 | 1
Urogenital (Renal and urinary disorders) | 0 | 1
Stomach cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Respiratory problems post-op; has COPD (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Antibiotics given imm post-op (General disorders) | 0 | 1 — Unknown if this was related to infection or other condition. No further information available.
2 units of blood given post-op (Blood and lymphatic system disorders) | 0 | 1
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Fall - soft tissue injury (General disorders) | 1 | 0
Hernia (General disorders) | 1 | 0
Non-traumatic bruising (General disorders) | 1 | 0
Needs scar revised (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No